CLINICAL TRIAL: NCT02021201
Title: The Effect of Sertindole and Risperidone on Endophenotypic Markers of Schizophrenia, a Comparative Study
Brief Title: The Effect of Sertindole and Risperidone on Endophenotypic Markers of Schizophrenia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No suitable patients could be recruited in the available time period
Sponsor: Birte Glenthoj (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor-Investigator, Birte Glenthoj, Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-A-2008-062
Record Dates: First submitted 2011-09-19; First posted 2013-12-27 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; sertindole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients with schizophrenia will be treated with risperidone or sertindole for a period of 10 weeks, after which they will cross-over for an additional treatment of 10 weeks with the other compound
  Interventions: Drug: risperidone; Drug: Sertindole
- 2 (Experimental): Patients with schizophrenia will be treated with risperidone or sertindole for a period of 10 weeks, after which they will cross-over for an additional treatment of 10 weeks with the other compound
  Interventions: Drug: risperidone; Drug: Sertindole

INTERVENTIONS:
Drug: risperidone — Patients with schizophrenia will be treated for 10 weeks treatment with risperidone
  Other Names: Risperdal
Drug: Sertindole — Patients with schizophrenia will be treated for 10 weeks treatment with serindole
  Other Names: Serdolect

SUMMARY:
This comparison is made between the effects of sertindole and risperidone on vulnerability indicators in schizophrenia. More specifically: the effects of these two antipsychotic compounds on basic processing of incoming information is studied. The investigators expect that the newer antipsychotic sertindole to be more effective in restoring information processing in schizophrenia patients than risperidone.

DETAILED DESCRIPTION:
The study is has a so-called double blind, randomized - yet balanced - cross-over design, in which 24 male patients with schizophrenia are included. After inclusion in the study, patients will be assessed in a test-battery, in which psychophysiological parameters of their basic information capabilities are quantified. Following this, the patients will be treated with either risperidone or sertindole for a period of 10 weeks, after which they will cross-over to the other treatment (the order of treatments is randomized (and balanced)). The battery of tests is repeated after the first and second treatment period. In addition, a second test-battery will be performed at these follow-up intervals, to assess neuropsychological parameters of information processing. To evaluate the extend of the treatment effects, the patients will be matched (age, gender, parental socioeconomic status) to 24 healthy controls.

ELIGIBILITY:
Inclusion Criteria:

Healthy controls:

* matched by age (+/- 2 years), gender and parental socioeconomic status to patients with schizophrenia.
* age between 18-55 years
* male
* physically and mentally healthy and no daily intake of medicine
* no current substance abuse

Patients:

* patients who fulfill both ICD-10 and DSM IV diagnostic criteria for schizophrenia.
* age between 18-55 years
* male
* patients who need a change in their medication
* diagnosed with schizophrenia within the last 10 years
* not formerly treated with risperidone (Risperdal) or sertindole (Serdolect) where treatment was stopped because of side effects or lack of effect
* physically healthy
* no current substance abuse

Exclusion Criteria:

Controls:

* a history of mental illness in the first degree relatives
* hearing disabilities
* head injury accompanied by unconsciousness for more than 5 min.
* physical illness with a need of daily intake of medicine
* positive screening for drugs of abuse at baseline.

Patients:

* head injury accompanied by unconsciousness for more than 5 min.
* serious medical conditions (more specific: brain diseases and diseases which cause a daily intake of medicine, heart, liver or kidney diseases, diabetes and prolongation of the QTc-interval (or a family history of such) and patients with phenylketonuri)
* abuse of alcohol or medication/ narcotics during the last 6 months or positive screening for drugs of abuse at baseline.
* former treatment with risperidone (Risperdal) or sertindole (Serdolect) where treatment was stopped because of side effects or lack of effect
* hearing disability
* allergy towards the content in the medicine used in the study
* bradycardia (pulse under 50 beats per minute) and QTc>450 ms

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2008-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Psychophysiological parameters sensory gating | baseline, after ten weeks and after 20 weeks

SECONDARY OUTCOMES:
Psychophysiological parameters of selective attention | Baseline, 10 weeks and 20 weeks after treatment
Neurocognitive parameters of amongst others executive functioning, attention, and reaction time | 10 weeks and 20 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Birte Y Glenthoj, PhD, Study Director — Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen, Psychiatric Center Glostrup; Bob Oranje, PhD, Principal Investigator — Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen, Psychiatric Center Glostrup; Birgitte Fagerlund, PhD, Principal Investigator — Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen, Psychiatric Center Glostrup; Rita S Godske, MD, Principal Investigator — Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen, Psychiatric Center Glostrup
Locations (1):
- Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen, Psychiatric Center Glostrup, Glostrup Municipality, Denmark

REFERENCES:
- See also: Homepage of our organization — https://www.psykiatri-regionh.dk/cinsr/Pages/default.aspx